CLINICAL TRIAL: NCT04697732
Title: The Incidence of Intraoperative Awareness Under General Anesthesia in Adults: A Prospective, Multicenter Study
Brief Title: İntraoperative Awareness Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Bahattin Tuncali, Associate professor, MD, Baskent University Ankara Hospital
Other Study IDs: KA12/154
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: To Investigate the Incidence and Causes of Awareness During General Anesthesia; To Investigate the of Dreaming During Anesthesia; To Investigate the Intra-operative Experiences of Patients Who Report Awareness; To Investigate the Risk Factors That May be Associated With Awareness; To Analyze the Frequency of Posttraumatic Stress Disorder in Cases With Awareness and Possible Awareness; To Investigate the Risk Factors That May be Associated With Posttraumatic Stress Disorder
Keywords: intraoperative awareness; general anesthesia; dreaming; incidence
MeSH Terms: conditions — Intraoperative Awareness | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients age above 18 years: ASA I-IV adult patients over 18 years of age who will receive general anesthesia and are scheduled to be extubated postoperatively, who can give informed consent, have no known psychological or psychiatric problems, and who are suitable for postoperative follow-up.
  Interventions: Other: General anesthesia

INTERVENTIONS:
Other: General anesthesia — Following emergence from general anesthesia, patients will be evaluated at 4 different timepoints; (a) One hour after emergence, (b) Twenty four hour after emergence (c) One week after emergence (d) One month after emergence. The first interview will be made face-to-face in the recovery unit, and other interviews will be made by phone.
  Other Names: Modified Brice Interview

SUMMARY:
Intraoperative awareness which means the recall of experiences recorded in patients' memories during general anesthesia in the postoperative period is an important issue in anesthesia practice. The aims of this study are to investigate the incidence and causes of awareness during general anesthesia, incidence of dreaming during anesthesia, intra-operative experiences of patients who report awareness, the risk factors that may be associated with awareness, to analyze the frequency of posttraumatic stress disorder in cases with awareness and possible awareness, the risk factors that may be associated with PTSD in Turkish adults.

Adult patients will be evaluated 4 time following emergence (a) One hour after emergence, (b) Twenty four hour after emergence (c) One week after emergence (d) One month after emergence. The first interview will be made face-to-face in the recovery unit, and other interviews will be made by phone. Each interview will be conducted using the same structured interview (Brice Interview).

Descriptive statistics will be used to determine the incidence of awareness. χ2 test will be used for comparison between groups. Logistic regression will be used to determine the risk factors associated with awareness and PTSD.

We believe that this study will contribute to the prevention of the problem by determining the real frequency and causes of intraoperative awareness under general anesthesia, determining the experiences and results of patients, and analyzing the associated risk factors.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-IV adult patients who will receive general anesthesia and are scheduled to be extubated postoperatively,

Exclusion Criteria:

* ASA V patients
* Patients below 18 years of age,
* Patient who can not give informed consent,
* Patients who have known psychological or psychiatric problems,
* Patients who are not suitable for postoperative follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-IV adult patients above 18 years of age who will receive general anesthesia and are scheduled to be extubated postoperatively,
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-07-17 (Actual); Primary Completion 2022-07-17 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Brice interview | One hour after emergence
  This interview consists of 5 questions. Patients will be evaluated at 4 different timepoints following emergence. First interview will be made face-to-face in the recovery unit, and other interviews will be made by phone.
Modified Brice interview | Twenty four hour after emergence
  This interview consists of 5 questions. Patients will be evaluated at 4 different timepoints following emergence. First interview will be made face-to-face in the recovery unit, and other interviews will be made by phone.
Modified Brice interview | One week after emergence
  This interview consists of 5 questions. Patients will be evaluated at 4 different timepoints following emergence. First interview will be made face-to-face in the recovery unit, and other interviews will be made by phone.
Modified Brice interview | One month after emergence.
  This interview consists of 5 questions. Patients will be evaluated at 4 different timepoints following emergence. First interview will be made face-to-face in the recovery unit, and other interviews will be made by phone.

CONTACTS AND LOCATIONS:
Overall Officials: Bahattin Tuncali, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sebel PS, Bowdle TA, Ghoneim MM, Rampil IJ, Padilla RE, Gan TJ, Domino KB. The incidence of awareness during anesthesia: a multicenter United States study. Anesth Analg. 2004 Sep;99(3):833-839. doi: 10.1213/01.ANE.0000130261.90896.6C. PMID 15333419
- [Background] Sandin RH, Enlund G, Samuelsson P, Lennmarken C. Awareness during anaesthesia: a prospective case study. Lancet. 2000 Feb 26;355(9205):707-11. doi: 10.1016/S0140-6736(99)11010-9. PMID 10703802
- [Background] Moerman N, Bonke B, Oosting J. Awareness and recall during general anesthesia. Facts and feelings. Anesthesiology. 1993 Sep;79(3):454-64. doi: 10.1097/00000542-199309000-00007. PMID 8363069
- [Background] Ghoneim M. The trauma of awareness: history, clinical features, risk factors, and cost. Anesth Analg. 2010 Mar 1;110(3):666-7. doi: 10.1213/ANE.0b013e3181cb5dfa. No abstract available. PMID 20185645
- [Background] Lennmarken C, Bildfors K, Enlund G, Samuelsson P, Sandin R. Victims of awareness. Acta Anaesthesiol Scand. 2002 Mar;46(3):229-31. doi: 10.1034/j.1399-6576.2002.t01-1-460301.x. PMID 11939910
- [Background] Mashour GA. Posttraumatic stress disorder after intraoperative awareness and high-risk surgery. Anesth Analg. 2010 Mar 1;110(3):668-70. doi: 10.1213/ANE.0b013e3181c35926. No abstract available. PMID 20185646
- [Background] Bischoff P, Rundshagen I. Awareness under general anesthesia. Dtsch Arztebl Int. 2011 Jan;108(1-2):1-7. doi: 10.3238/arztebl.2011.0001. Epub 2011 Jan 10. PMID 21285993
- [Background] Errando CL, Perez-Caballero P, Gelb AW, Sigl JC. Methodology, human factors, and incidence of intraoperative awareness. Acta Anaesthesiol Scand. 2010 Jul;54(6):781-3. doi: 10.1111/j.1399-6576.2010.02216.x. No abstract available. PMID 20618162
- [Background] Enlund M, Hassan HG. Intraoperative awareness: detected by the structured Brice interview? Acta Anaesthesiol Scand. 2002 Apr;46(4):345-9. doi: 10.1034/j.1399-6576.2002.460402.x. PMID 11952430
- [Background] Kotsovolis G, Komninos G. Awareness during anesthesia: how sure can we be that the patient is sleeping indeed? Hippokratia. 2009 Apr;13(2):83-9. PMID 19561776
- [Background] American Society of Anesthesiologists Task Force on Intraoperative Awareness. Practice advisory for intraoperative awareness and brain function monitoring: a report by the american society of anesthesiologists task force on intraoperative awareness. Anesthesiology. 2006 Apr;104(4):847-64. doi: 10.1097/00000542-200604000-00031. No abstract available. PMID 16571982
- [Background] WINTERBOTTOM EH. Insufficient anaesthesia. Br Med J. 1950 Jan 28;1(4647):247. doi: 10.1136/bmj.1.4647.247-c. No abstract available. PMID 15404998
- [Background] Sandlin D. A closer look at bispectral index monitoring. J Perianesth Nurs. 2001 Dec;16(6):420-2. doi: 10.1053/jpan.2001.28748. PMID 11740782
- [Background] Ishizawa Y. Mechanisms of anesthetic actions and the brain. J Anesth. 2007;21(2):187-99. doi: 10.1007/s00540-006-0482-x. Epub 2007 May 30. PMID 17458649
- [Background] Domino KB, Posner KL, Caplan RA, Cheney FW. Awareness during anesthesia: a closed claims analysis. Anesthesiology. 1999 Apr;90(4):1053-61. doi: 10.1097/00000542-199904000-00019. PMID 10201677
- [Background] Xu L, Wu AS, Yue Y. The incidence of intra-operative awareness during general anesthesia in China: a multi-center observational study. Acta Anaesthesiol Scand. 2009 Aug;53(7):873-82. doi: 10.1111/j.1399-6576.2009.02016.x. Epub 2009 Jun 3. PMID 19496761
- [Background] Errando CL, Sigl JC, Robles M, Calabuig E, Garcia J, Arocas F, Higueras R, Del Rosario E, Lopez D, Peiro CM, Soriano JL, Chaves S, Gil F, Garcia-Aguado R. Awareness with recall during general anaesthesia: a prospective observational evaluation of 4001 patients. Br J Anaesth. 2008 Aug;101(2):178-85. doi: 10.1093/bja/aen144. Epub 2008 May 30. PMID 18515816
- [Background] Pollard RJ, Coyle JP, Gilbert RL, Beck JE. Intraoperative awareness in a regional medical system: a review of 3 years' data. Anesthesiology. 2007 Feb;106(2):269-74. doi: 10.1097/00000542-200702000-00014. PMID 17264720
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Ekman A, Lindholm ML, Lennmarken C, Sandin R. Reduction in the incidence of awareness using BIS monitoring. Acta Anaesthesiol Scand. 2004 Jan;48(1):20-6. doi: 10.1111/j.1399-6576.2004.00260.x. PMID 14674969
- [Background] Wennervirta J, Ranta SO, Hynynen M. Awareness and recall in outpatient anesthesia. Anesth Analg. 2002 Jul;95(1):72-7, table of contents. doi: 10.1097/00000539-200207000-00013. PMID 12088946
- [Background] Ranta SO, Laurila R, Saario J, Ali-Melkkila T, Hynynen M. Awareness with recall during general anesthesia: incidence and risk factors. Anesth Analg. 1998 May;86(5):1084-9. doi: 10.1097/00000539-199805000-00035. PMID 9585303
- [Background] Nordstrom O, Engstrom AM, Persson S, Sandin R. Incidence of awareness in total i.v. anaesthesia based on propofol, alfentanil and neuromuscular blockade. Acta Anaesthesiol Scand. 1997 Sep;41(8):978-84. doi: 10.1111/j.1399-6576.1997.tb04823.x. PMID 9311394
- [Background] Schwender D, Kunze-Kronawitter H, Dietrich P, Klasing S, Forst H, Madler C. Conscious awareness during general anaesthesia: patients' perceptions, emotions, cognition and reactions. Br J Anaesth. 1998 Feb;80(2):133-9. doi: 10.1093/bja/80.2.133. PMID 9602573
- [Background] Osterman JE, van der Kolk BA. Awareness during anesthesia and posttraumatic stress disorder. Gen Hosp Psychiatry. 1998 Sep;20(5):274-81. doi: 10.1016/s0163-8343(98)00035-8. PMID 9788027
- [Background] Forman S. Awareness during general anesthesia: Concepts and controversies. Periop Med and Pain 2006; 25: 211-218
- [Background] Leslie K, Davidson AJ. Awareness during anesthesia: a problem without solutions? Minerva Anestesiol. 2010 Aug;76(8):624-8. PMID 20661203